CLINICAL TRIAL: NCT02520479
Title: Phase 2 Trial of "Sandwich" Pegaspargase-CHOP Chemotherapy With Radiotherapy in Newly Diagnosed, Stage IE to IIE, Nasal Type, Extranodal Natural Killer/T-cell Lymphoma
Brief Title: "Sandwich" Chemotherapy With Radiotherapy in Newly Diagnosed, Stage IE to IIE, ENKTL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, wanghua, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK-SYSUCC
Record Dates: First submitted 2015-08-04; First posted 2015-08-11 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2016-10

CONDITIONS: Treatment Refusal
Keywords: extranodal natural killer/T-cell lymphoma; nasal type; radiotherapy; chemotherapy
MeSH Terms: conditions — Treatment Refusal | interventions — pegaspargase; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sandwich protocols (Experimental): sandwich protocols: Patients with newly diagnosed ENKTL is given 2 cycles of P-CHOP[cyclophosphamide(CTX), 750 mg/m2 day 1; vincristine(VCR), 1.4 mg/m2 day 1 (maximal dose 2 mg),adriamycin(ADM) 50 mg/m2 day 1; dexamethasone(DXM) 10 mg days 1-8; Pegaspargase 2500 international unit day 1] before radiotherapy(RT) and then two "consolidation" cycles after RT.
  Interventions: Drug: P-CHOP; Radiation: Radiotherapy

INTERVENTIONS:
Drug: P-CHOP — Two cycles of P-CHOP:cyclophosphamide, 750 mg/m2 day 1; vincristine,(maximal dose 2 mg),adriamycin , 50 mg/m2 day 1; dexamethasone,10mg days 1-8; Pegaspargase, 2500IU/m2 day 1 are given before radiotherapy
  Other Names: CTX, VCR, ADM , DXM, Pegaspargase
Radiation: Radiotherapy — Radiotherapy was scheduled after 2 cycles of P-CHOPregimen. Involved field radiotherapy(IFRT) is delivered using 6-Million electron Volts linear accelerator using 3-dimensional conformable treatment planning. The IFRT dose was 56 grays (Gy) in 28 fractions.
  Other Names: radiotherapy after induction chemotherapy
Drug: P-CHOP — Two "consolidation" cycles of P-CHOP are given after radiotherapy
  Other Names: CTX, VCR, ADM , DXM, Pegaspargase

SUMMARY:
A phase 2 study was conducted of "sandwich" protocols, with earlier RT after an initial 2 of P-CHOP (Pegaspargase, cyclophosphamide,vincristine, doxorubicin and dexamethasone ), followed by further two "consolidation" cycles,to explore the appropriate mode of combined modality therapy (CMT) in early stage ENKTL.

DETAILED DESCRIPTION:
The extranodal natural killer/T-cell lymphoma (ENKTL) shows high local or systemic failure rates when radiotherapy (RT) is taken as the primary treatment, suggesting a role for chemotherapy (CT) added to RT for this disease. However, the appropriate mode of combined modality therapy (CMT) has not been fully defined.We conducted a prospective phase II study of "Sandwich" Pegaspargase, cyclophosphamide,vincristine, doxorubicin and dexamethasone (P-CHOP) regimen in combination with radiotherapy.The "sandwich" protocols, refer to earlier RT after an initial 2 cycles of P-CHOP followed by further two "consolidation" cycles.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed ENKTL
* age:18-69years
* Ann Arbor stage IE,or stage IIE with cervical lymph node involvement
* at lease one measurable lesion
* receive no chemotherapy or radiotherapy before
* Eastern CooperativeOncology Group performance status of 0 to 2.
* Adequate hematologic function (eg, white blood cell ≥ 3×10e9/l,neutrophils count ≥1.5×10e9/L, and platelet count≥ 100×10e9/L),renal function (eg, serum creatinine≤1.5 mg/dL and creatinine clearance ≥50 mL minute), and hepatic function (e.g, total bilirubin≤ 2 times the upper limit of normal and aspartate and alanine transaminase levels ≤ 3 times the upper limit of normal)

Exclusion Criteria:

* mismatch the inclusion criteria
* systematic central nervous system involvement
* previous or concomitant malignancies and any coexisting medical problems that could cause poor compliance with the study protocol.
* primary lesion not from the upper respiratory

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-06; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
complete remission rate | every 4 weeks,up to completion of treatment(approximately 6 months)
  The criteria for the efficacy evaluation (complete remission) of the regimen is according to the following article.
  Cheson BD, Horning SJ, Coiffier B, et al. Report of an international workshop to standardize response criteria for non-Hodgkin's lymphomas. NCI Sponsored International Working Group. J Clin Oncol. 1999;17:1244

SECONDARY OUTCOMES:
progression free survival | up to end of follow-up-phase (approximately 3 years)
  time from the date of enrollment to date of disease progression, or death of any cause, or date of lost follow-up, whichever comes first
overall survival | up to end of follow-up-phase (approximately 3 years)
  time from the date of enrollment to date of death from any cause, or date of lost follow-up, whichever comes first.
Hematological and non-hematological safety as a measure of adverse events according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE) | up to end of follow-up-phase (approximately 3 years)
  including hematological safety and non-hematological safety. All the adverse events will be classified according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: minghuang hong, MD., Study Director — Clinical Research Center
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China